CLINICAL TRIAL: NCT04302298
Title: The Role of Virtual Reality in Orthopaedic Surgery Education: A Randomized Control Trial
Brief Title: The Role of Virtual Reality in Orthopaedic Surgery Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mark H Gonzalez, Professor and Department Chair of the Department of Orthopaedics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-0335
Record Dates: First submitted 2020-02-11; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Virtual Reality; Surgical Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Medical students will be recruited via an email which asks them to participate in the trial. Those who respond will be randomly assigned into the virtual reality or technique guide group, and thus know which group they are a part of. They will be randomly assigned into these groups using a number generator of 1 or 2 for the virtual reality and technique guide group, respectively. An equal amount of participants will be allocated to each group.
  Following completion of the experiment, the attending physician evaluating their performance will be blinded to which group they were in as well as the gender of the participant to eliminate any bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): This group will go through the virtual reality simulation of a procedure prior to doing it on a plastic SawBone.
  Interventions: Device: Virtual Reality
- Technique Guide Group (No Intervention): This group will go be able to read through a technique guide on the procedure prior to doing it on a plastic SawBone. This is the current method of learning in surgical residencies.

INTERVENTIONS:
Device: Virtual Reality — A machine which immerses the participant in a simulated environment where they can perform a procedure.
  Arms: Virtual Reality Group

SUMMARY:
Virtual reality (VR) and augmented reality are becoming prominent in the medical sciences due to the increasing sophistication of VR technology and its improving haptics to simulate real-life situations. Previous medical VR studies focused on arthroscopic minimally-invasive procedures which often do not carry the risk of invasive procedures. OssoVR, an orthopedic surgery virtual reality company, has created a platform to run through different invasive orthopedic procedures prior to operating on a patient. Given that invasive procedures inherently carry more risk and variability than minimally invasive procedures, training tools to help with these operations are vital prior to performing on a patient. The research team will evaluate the face validity, transfer validity, and surgical recall of the orthopedic virtual reality software in an intramedullary (IM) tibial nail procedure. The research team will evaluate the simulation with medical students who have not had prior exposure to the procedure. Including medical students will allow for a larger sample size for more analysis. An IM tibial nail procedure is used in tibial fractures to help stabilize the fractured long bone via placement of a nail within the bone.

DETAILED DESCRIPTION:
Virtual reality has the potential to make a significant impact on medical education at both the medical student and resident level. OssoVR is one of the first companies that has produced functioning software for this niche student group. Medical students gain intimate knowledge regarding the musculoskeletal system helpful for the board exam and a unique insight into procedures they will see during clerkship. This offers them a larger potential to learn when seeing the procedure in the OR, and a view of orthopedic surgery they might not have if they decide to go into other specialties. Testing its efficacy on medical students will help reveal whether or not it may be helpful to have residents use virtual reality rather than reading a step-by-step guide, which is currently the norm for residents after observing the procedure performed by an attending. There is strong agreement in the literature that simulation technology should be a required part of orthopedic residence training (5) and that it improves resident surgical performance. The study was limited to medical students due to the limited number of orthopedic residents at UIC that have not seen an IM tibial nail procedure.

Objectives/Aims

Aim I. Test the procedural competence of the VR versus the step-by-step guide of IM tibial nail. I will have all of the students go through the procedure on SawBones separately. SawBones are artificial bones used to help train orthopedic students on how to perform a surgery prior to performing the surgery. To ensure blinding, Dr. Gonzalez evaluate their performance as he is a professional in orthopedic surgery and has the appropriate background for proper evaluation of accuracy. He will evaluate their time to complete the procedure, their accuracy in following the steps, and their OSATS score which is used to evaluate surgical technical skills.

Aim II. Evaluate how the students who completed the VR simulation felt regarding it. After going through the tibial nail simulation, the students will take a subjective survey regarding how they felt about the experience adapted from a current questionnaire used for virtual environment experiences .

ELIGIBILITY:
Inclusion Criteria:

* 1st or 2nd year medical students at University of Illinois at Chicago College of Medicine

Exclusion Criteria:

* if they had done or ever seen a tibial nail procedure in the past

Ages: 20 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Completion Rate | day 10-14
  Which participants completed the SawBones procedure

SECONDARY OUTCOMES:
Number of Steps Performed Correctly - Accuracy | Within 25 minutes
  How many steps did the subject follow as designated in the technique guide/virtual reality?
Time of Completion | up to 25 minutes
  How quickly did each participant complete the surgical procedure, if completed it all?

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Gonzalez, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago College of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No